CLINICAL TRIAL: NCT01362478
Title: Gene Promoter DNA Methylations and Their Relationships With Endophenotypes in Patients With Schizophrenia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Chun-Hsin Chen, Staff, Department of Psychiatry, Taipei Medical University WanFang Hospital
Other Study IDs: 99083
Record Dates: First submitted 2011-05-26; First posted 2011-05-30 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Schizophrenia
Keywords: schizophrenia; gene promoter; methylation; endophenotype; epigenetic
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Gene promoter DNA methylations
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case group
- Control group

SUMMARY:
Schizophrenia is a disabling mental disease affecting about 1% of the worldwide population. There is an overall heritability estimate of 68% for the underlying liability to schizophrenia. Molecular epigenetic studies can overcome the complexities of traditional genetic studies and provide a new framework for the search of etiological factors in schizophrenia.

DNA methylation provides an example of an epigenetic process that affects gene expression. Several postmortem experiments have found that increased DNA methylation at the glutamic acid decarboxylase (GAD67) and reelin promoter, and hypomethylation of membrane-bound catechol-O-methyltransferase (MB-COMT) promoter gene in prefrontal cortex of schizophrenia patients.

Because it is impossible to obtain brain tissue from schizophrenia patients clinically, the peripheral blood mononuclear cell (PBMC) can partly represent the brain gene expression. It has been reported to use PBMC as biomarkers for epigenetic abnormalities, such as histone acetylation and methylation, in schizophrenia. To the investigators best knowledge, gene promoter DNA methylation abnormalities in schizophrenia have been limited to postmortem study. It warrants to studying the DNA methylation using schizophrenia's PBMC.

Recently, endophenotype strategy has emerged as an important tool in understanding the genetic architecture of schizophrenia. Some cognitive functions, such as attention and working memory (WM), have been used as candidate endophenotypes for genetic studies in schizophrenia. Synchronized GABA neurotransmission in the dorsolateral prefrontal cortex is required for adequate attention and working memory, suggesting that impairments in GABA-mediated inhibition in the prefrontal cortex could contribute to the endophenotype presentations in schizophrenia.

DETAILED DESCRIPTION:
The study will be approved by Institutional Review Board of participated institutions before recruiting patients. We will recruit 60 patients with schizophrenia and 60 healthy control subjects after explaining the study goal and getting the informed consents.

We will evaluate the performance of continuous performance test (CPT) and working memory subset in Chinese version of WAIS-III in both case and control subjects. We will assay reelin, GAD, and MB-COMT gene promoter DNA methylation using methylation specific PCR (MSP) and quantify these gene expression using quantitative reverse transcription polymerase chain reaction (qRT-PCR).

Patients will be followed in one year and receive the same evaluation.

ELIGIBILITY:
Case

Inclusion Criteria:

* age 20-65 year-old
* fulfill DSM-IV criteria of schizophrenia

Exclusion Criteria:

* patients who are pregnant or have significant medical conditions
* unstable psychiatric features (e.g. suicidal), too agitation
* a history of substance abuse or drug addiction within the previous 6 months, with the exception of nicotine dependence.

Control

Inclusion Criteria:

* 20-65 year-old

Exclusion Criteria:

* to have major psychiatric disorder, such as schizophrenia, mood disorders, and substance use disorders, except nicotine
* to have family history of schizophrenia, mood disorders, and substance use disorders
* to have serious medical conditions

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: schizophrenia patients
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2011-08; Study Completion 2014-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Hsin Chen, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (2):
- Taiwan (2):
  - WanFang Hospital, Taipei Medical University, Taipei, Taiwan
  - Taipei Medical University - WanFang Hospital, Taipei